CLINICAL TRIAL: NCT02690740
Title: Titrated Quantitative Conjunctival Provocation Test (tqCPT): Standardization and Validation of a New Clinical Endpoint
Brief Title: Titrated Quantitative Conjunctival Provocation Test (tqCPT)
Acronym: tqCPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zentrums für Rhinologie und Allergologie Wiesbaden (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AZ_001_CPT
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Allergic Rhinitis
Keywords: titrated quantitative conjunctival provocation test
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): test/retest of a titrated quantitative CPT (TqCPT) with outcomes: CPT-scoring system and correlation with digital photo analysis.
  in all patients: 1 Arm = CPT test/re-test, no comparator
  No intervention of a new drug (CPT-solution registered (ALK- Abelló, Hørsholm, Denmark));
  Interventions: Other: (diagnostic) conjunctival provocation test with solution: ALK 100, 1.000, 10.000, 20.000, 50.000 and 100.000 SQ-U/ml

INTERVENTIONS:
Other: (diagnostic) conjunctival provocation test with solution: ALK 100, 1.000, 10.000, 20.000, 50.000 and 100.000 SQ-U/ml — see information in "arm/group descriptions"

SUMMARY:
The clinical relevance of an allergen-specific sensitization is proven e.g., by allergen challenge tests in clinical routine. Several protocols for different challenge tests such as nasal (NPT), bronchial (BPT) or conjunctival provocation test (CPT) have been proposed. Beneath others, the CPT is broadly used in both clinical trials and routine because of its feasibility.

However, there is no internationally harmonized standard regarding the clinical interpretation of CPT results as well as a lack of validation of a specific outcome score. Therefore, this trial aims to investigate and validate a new scoring system for CPT results in order to provide this test as a useful method in future clinical trials.

DETAILED DESCRIPTION:
Of 33 patients who had been initially screened, ten patients did not fulfill all of the inclusion criteria mentioned hereafter. Thus, 23 patients aged 18 to 67 years having a birch and/or grass pollen allergy were included in the analysis. The study is in line with the Declaration of Helsinki and is approved by the responsible ethics committee (FF 118/2012 (4 December 2012); Landesärztekammer Hessen, Frankfurt, Germany). All participating patients are informed of the nature and objectives of the study and signed an informed consent document.

The CPT is conducted using standardized and registered allergen extracts (ALK- Abelló, Hørsholm, Denmark). At the first visit, a titrated quantitative CPT (tqCPT) is performed according to a standardized protocol. In case of a positive test result, CPT-results are to be confirmed at a re-challenge one week later. The final CPT takes place 3 to 4 weeks after the 2nd (confirmatory) challenge for analyzing the primary objective of the trial: reproducibility of the CPT symptom score. Furthermore, objective evaluation of the clinical reactions after the tqCPT is documented using a MATLAB software program to calculate the degree of redness in percent. This is then correlated with the (subjective) main investigators' evaluations and with the external observer's evaluations.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe allergic rhinoconjunctivitis (ARC) symptoms in preceding two years -intake of anti-allergic medication in the preceding two years -positive test result in skin prick test (SPT) (wheal size at least 3 mm larger than the negative control). -
* retrospective global symptoms score (≥5 out of 12)

Exclusion Criteria:

* acute diseases of the eye or of the nose/nasal sinuses,
* persistent allergy
* intake of concomitant (antiallergic) medication prior to CPT-challenges
* CPT score ≥3 during the examination of the control (non-challenged eye) at baseline

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
total conjunctival symptoms provoked by conjunctival provocation test (CPT) at two consecutive settings | baseline and re-challenge after 3-4 weeks
  Total Conjunctival symptoms (itching (0-3), irritation (0-3), tearing (0-3), redness (0-3)) provoked by a conjunctival provocation test (CPT) were evaluated and categorized on a 4 point Likert-Scale (Total Score = 0-12 points)) at a first setting and then again after a rechallenge after an interval of 3-4 weeks. Changes of Total score values (0-12 points) of both settings were calculated using the the Pearson and Spearman correlation coefficients.

SECONDARY OUTCOMES:
Conjunctival redness score (0-3) provoked by conjunctival provocation test (CPT) at two consecutive settings. | baseline and re-challenge after 3-4 weeks
  Conjunctival redness provoked by a conjunctival provocation test (CPT) was evaluated and categorized on a 4 point Likert-Scale (0-3) at a first setting and then again after a rechallenge after an interval of 3-4 weeks. Changes of the conjunctival redness score of both settings were calculated using the the Pearson and Spearman correlation coefficients.
difference in the degree of conjunctival redness provoked by conjunctival provocation test (CPT) at two consecutive settings as assessed by digital photo analysis | baseline and re-challenge after 3-4 weeks
  Degree of conjunctival redness provoked by conjunctival provocation test (CPT) was assessed by digital photo analysis at a first setting and then after a rechallenge of 3-4 weeks. The percent change in the redness area was determined by a special software program.
Correlation of the degree of conjunctival redness as assessed by digital photo analysis with the conjunctival redness score evaluated and categorized on a 4 point Likert-Scale (0-3) provoked by a conjunctival provocation test (CPT). | baseline and re-challenge after 3-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pfaar, Prof.Dr., Principal Investigator — Allergy Center Wiesbaden, Germany; Ludger Klimek, Prof. Dr., Study Director — Allergy Center Wiesbaden, Germany; Dan Philipp Claßen, Study Chair — Allergy Center Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfaar O, Classen DP, Astvatsatourov A, Klimek L, Mosges R. Reliability of a New Symptom Score in a Titrated Quantitative Conjunctival Provocation Test Supported by an Objective Photodocumentation. Int Arch Allergy Immunol. 2018;176(3-4):215-224. doi: 10.1159/000487884. Epub 2018 May 16. PMID 29768274